CLINICAL TRIAL: NCT00590018
Title: Corticosteroids in Postoperative Critically Ill Neonates With Low Cardiac Output Syndrome With Congenital Heart Disease
Acronym: Corti
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Heather Dickerson, MD, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: H-12030
Record Dates: First submitted 2007-12-28; First posted 2008-01-10 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Cardiac Output, Low
Keywords: Congenital heart disease.; Low cardiac output syndrome.; Corticosteroids.; Hydrocortisone.; Blood pressure.; Inotropes.
MeSH Terms: conditions — Cardiac Output, Low; Heart Defects, Congenital | interventions — Hydrocortisone; Adrenal Cortex Hormones; Steroids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Subjects in this arm will receive a 5 day tapering course of hydrocortisone.
  Interventions: Drug: Hydrocortisone
- 2 (Placebo Comparator): Subjects in this arm will receive 5 days of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrocortisone — Hydrocortisone taper (100mg/m2/day --> 25mg/m2/day) over 5 days intravenously.
  Other Names: Corticosteroids.; Steroids.
  Arms: 1
Drug: Placebo — Placebo for 5 days intravenously.
  Arms: 2

SUMMARY:
Babies having heart surgery often have problems after surgery with their blood pressure and getting enough blood to their bodies. To treat this they require medicines to keep their blood pressure high enough to get blood to their bodies. The side effects of these medicines include fast heart rates and increasing the amount of work the heart has to do. Corticosteroids are made by the body and help to use the energy in the food people eat, control the chemicals in their blood and maintain their blood pressure. Corticosteroids made by the body may be decreased in patients that have major surgery. Corticosteroids help to increase blood pressure and can decrease the amount of blood pressure medicines a patient requires. Corticosteroids have been shown to increase blood pressure in patients with bacterial infections and in very small, premature babies but have only been studied in a few babies who have had heart surgery. The way corticosteroids work is unknown but may involve decreasing the body's response to being on a heart-lung machine or give steroids not being made by the patient.

Corticosteroids have been shown to be helpful in treating many diseases. The purpose of this study is to look at the effects of corticosteroids in babies who have had heart surgery and need blood pressure medicines in the intensive care unit after surgery. Our idea is that getting corticosteroids will allow us to decrease the amount of blood pressure medicines each patient needs and improve how they do after surgery. We also plan to do blood tests to help determine how the corticosteroids are working.

It will be randomly determined if the subject receives corticosteroids or salt water. The subject will receive a corticosteroid or salt water once a day for five days. Their vital signs will be monitored, especially blood pressure and their need for medicines to increase their blood pressure. Blood work will also be obtained to determine their body's ability to make steroids.

DETAILED DESCRIPTION:
The study will be prospective. Patients who meet entry criteria will be randomized to receive corticosteroids versus placebo. Randomization will take into account biventricular versus univentricular repairs/palliations and whether the patients received intraoperative steroids. Patients will be compared with matched controls based on: diagnosis, +/- intraoperative steroids/phenoxybenzamine, cardiopulmonary bypass/cross clamp/circulatory arrest times and inotrope requirements. Those in the treatment arm will be dosed with hydrocortisone - stress dose (100mg/m2/dose daily x2, then taper with two days at half the original dose and one day at one quarter of the original dose) and then the steroids will be discontinued. Outcome data will include: heart rate, blood pressure, mixed venous oxygen saturation to assess cardiac output, blood cultures/infection/antibiotics (antibiotics as deemed necessary by the primary cardiologist), +/- gastrointestinal bleeding, time to discontinuing inotropic agents, time to extubation, length of intensive care unit admission and survival. Laboratory studies will be assessed before and 24 hours after the institution of steroids. The following labs are standard of care in the unit and will be assessed: glucose, electrolytes, blood urea nitrogen/creatinine, complete blood counts, lactate, arterial blood gases, cultures and stool guaiac. The following labs will be assessed in addition to regular monitoring: cortisol, adrenocorticotropin hormone and C reactive protein.

ELIGIBILITY:
Inclusion Criteria:

* Age < 1 month
* Postoperative
* Inotrope score > 20 x > 4 hrs [epinephrine: (mcg/kg/min) x 100 + norepinephrine: (mcg/kg/min) x 100 + phenylephrine: (mcg/kg/min) x 100 + vasopressin: (units/kg/hr) x 100 + milrinone: (mcg/kg/min) x 15 + dopamine: (mcg/kg/min) x 1 + dobutamine: (mcg/kg/min) x 1 + calcium chloride: (mg/kg/hr) x 1]

Exclusion Criteria:

* Age > 1 month
* Documented sepsis
* Preoperative use of steroids > 1 wk

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2003-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather A Dickerson, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Suominen PK, Dickerson HA, Moffett BS, Ranta SO, Mott AR, Price JF, Heinle JS, McKenzie ED, Fraser CD Jr, Chang AC. Hemodynamic effects of rescue protocol hydrocortisone in neonates with low cardiac output syndrome after cardiac surgery. Pediatr Crit Care Med. 2005 Nov;6(6):655-9. doi: 10.1097/01.pcc.0000185487.69215.29. PMID 16276331
- [Derived] Gibbison B, Villalobos Lizardi JC, Aviles Martinez KI, Fudulu DP, Medina Andrade MA, Perez-Gaxiola G, Schadenberg AW, Stoica SC, Lightman SL, Angelini GD, Reeves BC. Prophylactic corticosteroids for paediatric heart surgery with cardiopulmonary bypass. Cochrane Database Syst Rev. 2020 Oct 12;10(10):CD013101. doi: 10.1002/14651858.CD013101.pub2. PMID 33045104

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydrocortisone: Subjects in this arm will receive a 5 day tapering course of hydrocortisone. Hydrocortisone: Hydrocortisone taper (100mg/m2/day --> 25mg/m2/day) over 5 days intravenously.
- Placebo: Subjects in this arm will receive 5 days of placebo. Placebo: Placebo for 5 days intravenously.
Period: Overall Study
Arm/Group | Hydrocortisone | Placebo
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrocortisone | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 9 | 18
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 10 (10.58) | 7 (4.12) | 8.5 (7.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18
Inotrope score [Mean (Standard Deviation); unit: units on a scale] — Inotrope score: epinephrine (mcg/kg/min x 100) + norepinephrine (mcg/kg/min x 100) + phenylephrine (mcg/kg/min x 100) + dopamine (mcg/kg/min x1) + dobutamine (mcg/kg/min x 1) + milrinone (mcg/kg/min x15). The higher the score the higher the inotrope requirements and generally the sicker the patient. Minimum would be 0. Maximum would be 85.
  units on a scale | 23.46 (3.79) | 22.11 (2.31) | 22.78 (3.12)

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure.
Description: Change in mean blood pressure recorded prior to (15 minutes prior to study drug) and subsequent to medication/placebo administration (at 2 days post drug administration).
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 9 | 9
mmHg | 6 (7.86) | 5.89 (9.24)

2. Secondary Outcome: Change in Inotrope Score. This is the Change in the Inotrope Score Between 15 Minutes Prior to Drug Administration and at 2 Days After Drug Administration.
Description: Inotrope score: epinephrine (mcg/kg/min x 100) + norepinephrine (mcg/kg/min x 100) + phenylephrine (mcg/kg/min x 100) + dopamine (mcg/kg/min x1) + dobutamine (mcg/kg/min x 1) + milrinone (mcg/kg/min x15). A lower inotrope score is better with the minimum being 0 and the maximum being 85.
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 9 | 9
units on a scale | 8.83 (9.61) | 7.17 (4.8)

ADVERSE EVENTS:
Time Frame: Duration of the the admission time in the intensive care unit and hospital stay (duration of the study). This time period averaged 45 days.
Arm/Group | Hydrocortisone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocortisone (N=9) | Placebo (N=9)
Death (Cardiac disorders) | 0 (0) | 1 (1) — Death likely underlying heart disease - worsening function & arrhythmias. Study drug 9/20/04-9/24/04. No infections or bleeding. Weaned from inotropes after study drug. Deteriorated subsequently. Cleared by data safety monitoring board.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes